CLINICAL TRIAL: NCT06225505
Title: Early Detection of Triple Negative Breast Cancer Relapse: a Clinical Utility Phase II Trial
Brief Title: Early Detection of Triple Negative Breast Cancer Relapse (CUPCAKE)
Acronym: CUPCAKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: National Research Agency, France (Other); Roche Pharma AG (Industry); Personalis Inc. (Industry); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IC 2022-02
Record Dates: First submitted 2023-12-12; First posted 2024-01-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple negative breast cancer; 68Ga-FAPI-46; ctDNA
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: CUPCAKE is a randomized, non-comparative, multicenter, proof-of-concept phase II trial, using the Trials within Cohorts concept to assess the clinical utility of ctDNA monitoring combined with 68Ga-FAPI-46-PET-CT imaging upon ctDNA detection for the surveillance of patients with a non-metastatic TNBC at high risk of relapse.
  68Ga-FAPI-46 is the radiopharmaceutical product. There is no study treatment (standard of Care).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Upon detection of ctDNA during Step1, patients will be centrally assigned to the control or the experimental arm (1:1) using the eCRF.
  Randomization will be stratified by RCB score (I/II vs. III/NA because no neoadjuvant chemotherapy) and by time to molecular relapse (< 12 months vs. ≥ 12 months between surgery and molecular relapse).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): In the experimental arm, patients and their treating physician will be made aware of the molecular relapse (positive ctDNA detection results) in study steps 1 (ctDNA monitoring). To locate metastatic deposits, patients will be offered to undergo a whole-body imaging with 18F-FDG PET-CT and 68Ga-FAPI-46-PET-CT, in addition to any other workup considered as relevant by their treating physician.
  Interventions: Diagnostic Test: ctDNA monitoring; Diagnostic Test: 68Ga-FAPI-46-PET-CT
- Control arm (Sham Comparator): In the control arm, patients and their treating physician will not be made aware of the molecular relapse and will continue the standard surveillance with repeated ctDNA test every 4 months (blinded). ). At the time of the clinical/radiological diagnosis of relapse, similar procedures will be performed (18F-FDG PET-CT, 68Ga-FAPI-46-PET-CT, and tumor genetic landscape assessment by ctDNA analysis).
  Interventions: Diagnostic Test: ctDNA monitoring; Diagnostic Test: 68Ga-FAPI-46-PET-CT

INTERVENTIONS:
Diagnostic Test: ctDNA monitoring — For each patient included, a ctDNA detection assay will be performed in blood samples every 4 months, while extra-plasma will be banked. ctDNA results will be available with a turnaround time of less than 3 weeks. When negative, ctDNA detection results will not be disclosed to patients nor clinicians.
Diagnostic Test: 68Ga-FAPI-46-PET-CT — ). To locate metastatic deposits, patients will be offered to undergo a whole-body imaging with 18F-FDG PET-CT and 68Ga-FAPI-46-PET-CT, in addition to any other workup considered as relevant by their treating physician.

SUMMARY:
CUPCAKE is a randomized, non-comparative, multicenter, proof-of-concept phase II trial, using the Trials within Cohorts concept(1) to assess the clinical utility of ctDNA monitoring combined with 68Ga-FAPI-46-PET-CT imaging upon ctDNA detection for the surveillance of patients with a non-metastatic TNBC at high risk of relapse.

The study has two steps. In Step 1, patients who have completed the treatments for a localized TNBC will undergo ctDNA monitoring every ~4 months (± 2 weeks). In Step 2, patients for whom ctDNA will be detected will then be randomized between an observation arm, in which monitoring will continue until the detection of a clinical relapse, and an experimental arm, in which the ctDNA detection will be revealed to both the patient and the clinician: patients will then undergo a 18F-FDG PET-CT and a 68Ga-FAPI-46-PET-CT, in addition to whatever workup the investigator will deem necessary.

DETAILED DESCRIPTION:
The CUPCAKE trial will follow the Trials within Cohorts (TwiCs) approach. Non-metastatic TNBC patients at high risk of relapse will be included, after having signed a written informed consent, in a cohort allowing them to be followed by ctDNA monitoring every 4 months.

For each patient included, a ctDNA detection assay will be performed in blood samples every 4 months for a maximum of 24 months, while extra-plasma will be banked. ctDNA results will be available with a turnaround time of less than 3 weeks. When negative, ctDNA detection results will not be disclosed to patients nor clinicians.

First line therapy will not be started until a metastatic relapse has been found by imagining: no treatment will be started in the sole basis of a positive ctDNA test.

If, at any timepoint, ctDNA is detected (molecular relapse), patients will be randomized in a 1:1 ratio.

* In the experimental arm, patients and their treating physician will be made aware of the molecular relapse (positive ctDNA detection results). To locate metastatic deposits, patients will be offered to undergo a whole-body imaging with 18F-FDG PET-CT and 68Ga-FAPI-46-PET-CT, in addition to any other workup considered as relevant by their treating physician. If/when a clinical/radiological relapse is observed, the patient performance status will be registered (secondary objective) and systemic or local treatments will be decided by physicians. These treatments could be informed by the genetic landscape of the relapse, assessed by ctDNA.
* In the control arm, patients and their treating physician will not be made aware of the molecular relapse and will continue the standard surveillance with repeated ctDNA test every 4 months (blinded) for a maximum of 24 months from enrolement in the study. At the time of the clinical/radiological diagnosis of relapse, similar procedures will be performed (18F-FDG PET-CT, 68Ga-FAPI-46-PET-CT, and tumor genetic landscape assessment by ctDNA analysis).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed a written informed consent before inclusion
2. Patients must be female ≥ 18 years old
3. Patients diagnosed with a non-metastatic TNBC (ER & PR <10%, HER2- per ASCO/CAP guidelines). Patients must have been previously evaluated by a 18F-FDG PET-CT or a bone scintigraphy combined with a thorax, abdomen and pelvis CT scan with contrast
4. Patients who have undergone surgery with curative intent for their non-metastatic TNBC. Surgery must have been performed between 3 to 9 months before inclusion. Patients must have initiated their adjuvant therapy, whenever indicated, since at least 12 weeks. For patients receiving an experimental adjuvant treatment in a clinical trial, any intervention planned as part of this trial must be completed before inclusion.
5. High-risk primary tumor, defined as:

   1. Lack of pathological complete response after neoadjuvant chemotherapy (RCB I, II or III; RCB I being capped to a maximum of 30% of included patients) OR, in the absence of neoadjuvant chemotherapy,
   2. Stage IIB-III (i.e., T2N1, any T3-T4, any N2-3) OR
   3. Any loco-regional relapse occurring after a prior ipsilateral, curatively treated TNBC
6. No sign of local or distant relapse, as per investigator assessment
7. Performance status < 2
8. Available FFPE tumor block with > 10% cellularity or 11 tumor sections with >10% cellularity
9. Patient able to comply with protocol requirements
10. Patients covered by a health insurance

Exclusion Criteria:

1. Any uncontrolled disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding or any other medical condition that, in the opinion of the investigator, interferes with the trial procedures
2. Male participants
3. Patients with altered mental status or psychiatric disorder that, in the opinion of the investigator, would preclude a valid patient informed consent.
4. Patients who have difficulty undergoing trial procedures for geographic, social or psychological reasons
5. Person deprived of liberty or under guardianship
6. History of another primary malignancy except for the following :

   1. Basal cell carcinoma or any in situ carcinoma treated with curative intent
   2. Any stage I-II malignancy treated with curative intent with no evidence of active disease in the last five years
7. For step #2 (randomization after ctDNA detection): clinical/radiological metastatic relapse before the detection of the molecular relapse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2031-08-03 (Estimated); Study Completion 2031-08-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 36 months
  OS rate for the main analysis (primary endpoint) is defined as the percentage of patients still alive 36 months after the randomization. If the patient is not present at the 36th month visit, survival data may be obtained by other means, such as telephone contact with the patient, his family, his current physician, or consulting local death registries.
  A non-comparative analysis will be conducted in the experimental arm, and the control arm will serve as reference.

SECONDARY OUTCOMES:
Number of metastatic sites at the time of the clinical/radiological relapse. | Clinical/radiological relapse up to 36 months
  The number of metastatic sites upon clinical/radiological relapse will be defined post-hoc by the Adjudication Committee as the number of organs or systems in which metastases are detected at the time of the clinical/radiological relapse, among the following propositions: lymph nodes, bones, liver, lungs, central nervous system/meninges, peritoneum, others.
Recurrence-free survival | Clinical/radiological relapse up to 36 months
  RFS [recurrence-free survival], defined as the time from randomization to clinical/radiological relapse or death; PFS [progression-free survival], defined as the time from randomization to the first progression or death occurring after clinical/radiological relapse; 1L-PFS [first line PFS], defined as the time from clinical/radiological relapse to first progression or death ; 2L-PFS [second line PFS], defined as the time from first to second progression or death; progression being defined per RECIST criteria.
Overall response rate | 12 months
  Best ORR is defined as the proportion of patients with a complete response (CR) or partial response (PR) based on local investigator assessment according to RECIST 1.1, until first progression or last tumor assessment in the absence of progression. ORR will be reported with its 95% confidence interval by arm.
Overal Survival | Up to 36 months
  Overall Survival is defined as the time between randomization and death.
Performance Status Scale | Clinical/radiological relapse up to 36 months
  Proportion of patients presenting with an altered general condition (PS ≥2) at first evidence of clinical or radiological relapse.
  The population of interest consists in randomized patients.
EORTC Core Quality of Life questionnaire (EORTC-QLQ-C30) with the QLQ-BR42 module | Clinical/radiological relapse up to 36 months
  The EORTC-QLQ-C30 questionnaire with the QLQ-BR42 is used to report health-related QoL in all included patients. Summary statistics of the scores for all functional/symptom scales will be calculated at each assessment time point, according to the scoring procedure recommended by the EORTC.
  All of the scales and single item measures range in score from 0 to 100. A high score for the functional scales and functional single items represents a high/healthy level of functioning, whereas a high score for the symptom scales and symptom item represents a high level of symptomatology or problems.
5-level EQ-5D version (EQ-5D-5L) | Clinical/radiological relapse up to 24 months
  y. Each state is referred to in terms of a 5 digit code. For example, state 11111 indicates no problems on any of the 5 dimensions, while state 12345 indicates no problems with mobility, slight problems with washing or dressing, moderate problems with doing usual activities, severe pain or discomfort and extreme anxiety or depression. A completely healthy patient would have a score of 11111. This 5-digit number can be converted into a score using a special algorithm that is not publicly available. This point value is called the EQ-5D-5L Index and represents the patient's health status.
Proportion of patients receiving local treatment for oligometastatic disease | 36 months
  Proportion of patients receiving local treatment for oligometastatic disease

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément BIDARD, Principal Investigator — Institut Curie
Locations (13):
- France (13):
  - Sainte-Catherine Institut du Caner Avignon-Provence, Avignon
  - Institut Bergonié, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut du cancer de Montpellier, Montpellier
  - CHU Nîmes, Nîmes
  - Hôpital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - Centre Eugène Marquis, Rennes
  - Institut Curie, Saint-Cloud
  - ONCOPOLE Claudius Regaud, Toulouse
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accrodance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).